CLINICAL TRIAL: NCT04816630
Title: Feasibility Study to Evaluate Performance of MDW and Other Hematology Parameters for Identification of COVID-19 Disease and Clinical Progression in Adult Hospitalized Patients - Washington University
Brief Title: Feasibility Study of Hematology Parameters in COVID-19 Disease
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C71934
Record Dates: First submitted 2021-03-15; First posted 2021-03-25 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Covid19; Sepsis; Adults; Emergency Department
MeSH Terms: conditions — COVID-19; Sepsis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CBC-Diff Monocyte Volume Width Distribution: Monocyte Distribution Width [MDW] is part of the CBC with Differential. No intervention
  Interventions: Device: CBC-Diff Monocyte Volume Width Distribution

INTERVENTIONS:
Device: CBC-Diff Monocyte Volume Width Distribution — MDW is part of the CBC-Diff and will be collected but not reported to the physician. MDW will not impact standard of care.

SUMMARY:
The purpose of this study is to evaluate the potential for MDW and other CPD parameters (measured with CBC-DIFF) to identify COVID-19 diseased adult individuals presenting to the hospital with symptoms suggestive of COVID-19 or respiratory infection and whose standard of care includes CBC-DIFF and microbial testing.

DETAILED DESCRIPTION:
The objective of this study is to evaluate MDW and/or combination(s) of hematology parameters that best identify patients with COVID-19 disease who tested SAR-CoV-2 positive by standard of care (SOC) COVID-19 testing.

A feasibility study of consecutive adult patients who presented to the hospital with symptoms suggestive of COVID-19 or respiratory infection and whose standard of care testing involves a CBC-DIFF and microbial testing including RT-PCR testing for SARS-CoV-2 will be enrolled. This study will evaluate MDW and other CPD parameters performance in COVID-19 patients and the ability of MDW to identify RT-PCR positive COVID-19 patients as well as potential added value to RT-PCR tests of MDW. A minimum of 50 COVID-19 positive and 150 COVID-19 negative patients meeting inclusion criteria will be evaluated. Patients with symptoms suggestive of COVID-19 and who have RT-PCR test samples drawn will be retested on the DxH900 hematology analyzer to capture baseline MDW results. In addition, a retrospective data extraction will be performed for those patient samples tested during the Post Market study during the COVID-19 pandemic that meet the revised study population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients [18-89 years of age]
* Present to the Emergency Department
* With symptoms suggestive of COVID-19 or respiratory infection
* Whose assessment includes CBC-Diff and RT-PCR testing

Exclusion Criteria:

* Pregnancy
* Prisoners
* <18 years of age
* >89 years of age
* Previously evaluated in this study
* No RT-PCR testing
* Sample age >2 hours from time of draw
* Instrument flags, including vote outs and review flags for the MDW parameter
* Samples stored in refrigerated temperatures

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult (18 to 89 years) of all race and ethnicities presenting to the emergency department with symptoms suggestive of COVID-19 or respiratory infection and whose assessment includes a CBC-DIFF and microbial testing to include RT-PCR for SARS-CoV-2
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
COVID-19 diseased patients | Within 12 hours from presentation to the emergency department
  MDW's ability to identify COVID-19 negative versus COVID-19 positive patients using RT-PCR

SECONDARY OUTCOMES:
COVID-19 diseased patients diagnosed clinically | Within 12 hours from presentation to the emergency department
  MDW's ability to identify COVID-19 diseased patients versus site's COVID-19 diagnosis, including those that were RT-PCR negative

OTHER OUTCOMES:
Initial Disposition: Hospitalization | Within 12 hours from presentation to the emergency department
  MDW's ability to identify COVID-19 patients who require hospitalization
Initial Disposition: ICU Admission | Within 12 hours from presentation to the emergency department
  MDW's ability to identify COVID-19 patients who require treatment in the intensive care unit
Increased Respiratory Requirements such as Non-invasive and Invasive Mechanical Interventions | Within 72 hours from presentation to the emergency department
  MDW's ability to identify COVID-19 patients upon emergency department that may require increased respiratory requirements in 72 hours from presentation
COVID-19 Severity | Within 12 hours from presentation to the emergency department
  MDW's ability to identify COVID-19 patient severity [mild, moderate, severe and critical]

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Osborn, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No